CLINICAL TRIAL: NCT05273489
Title: Effect of Chemotherapy and Tumor Clearance in Hepatic Resections for Colorectal Liver Metastases. A Single-centre Cohort Study
Brief Title: Chemotherapy and Tumor Clearance in Hepatic Resections for Colorectal Liver Metastases.
Status: Completed | Type: Observational
Sponsor: Hospital Maciel (Other)
Collaborators: University of Adelaide (Other)
Responsible Party: Principal Investigator, Mauro Andres Perdomo, MD, MHA, MD, General Surgeon, Hospital Maciel
Other Study IDs: CRLM1
Record Dates: First submitted 2022-02-24; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer Metastatic; Liver Metastases
MeSH Terms: interventions — Hepatectomy; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Hepatectomy — Neoadjuvant treatment
  Other Names: Chemotherapy

SUMMARY:
Retrospective analysis of a prospectively collected database of 170 patients between 2004 and 2020, who underwent liver resections for CRLM (colorectal liver metastases) at The Queen Elizabeth Hospital trying to determine rates and patterns of recurrence following liver resections for CRLM and concurrently, characterise clinical, pathological and treatment-related factors that could function as predictors of recurrence or survival, particularly neoadjuvant chemotherapy and tumour clearance.

DETAILED DESCRIPTION:
This is a descriptive, observational study with retrospective analysis of a prospectively collated database. This database included all patients who underwent curative hepatic resections for CRLM (colorectal liver metastases) at The Queen Elizabeth Hospital (Adelaide, Australia) between December 2004 and October 2020.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a liver resection for CRLM at The Queen Elizabeth Hospital between December 2004 to September 2020

Exclusion Criteria:

* Patients whose procedures were abandoned due to unresectable tumour burden

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Australian citizens (most of them locals) treated at The Queen Elizabeth Hospital, Adelaide, SA.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Recurrence | From surgery to recurrence, up to 16 years
  Recurrence rate
Survival | From surgery to death or end of the study, up to 16 years
  up to16 years

SECONDARY OUTCOMES:
Resection margins | From surgery to death or end of the study, up to 16 years
  Resection margins of the liver resection
Neoadjuvant Chemotherapy | From surgery to death or end of the study, up to 16 years
  Neoadjuvant Chemotherapy (yes or not)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro A Perdomo, MD, MHA, Principal Investigator — Assitant Professor at Clinica Quirurgica 3. Universidad de la Republica. Monteviedo, Uruguay

IPD SHARING:
Plan to Share IPD: No
Data could be provided on reasonable request

DOCUMENTS (1):
  • Study Protocol (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT05273489/Prot_000.pdf